CLINICAL TRIAL: NCT01701050
Title: COMETI Phase 2: Characterization of Circulating Tumor Cells (CTC) From Patients With Metastatic Breast Cancer Using the CTC-Endocrine Therapy Index
Brief Title: Characterization of Circulating Tumor Cells (CTC) From Patients With Metastatic Breast Cancer Using the CTC-Endocrine Therapy Index
Acronym: COMETI P2
Status: Completed | Type: Observational
Sponsor: Janssen Diagnostics, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: COMETI-P2-2012
Record Dates: First submitted 2012-10-01; First posted 2012-10-04 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Metastatic Breast Cancer
Keywords: circulating tumor cells; CTC; metastatic breast cancer; endocrine therapy; hormone therapy
MeSH Terms: conditions — Breast Neoplasms; Neoplastic Cells, Circulating | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cartridges containing Circulating Tumor Cells (isolated by CellSearch) as well as primary and/or metastatic tumor tissue (blocks or slides).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Blood collection: Female patients 18 years or older with estrogen receptor (ER) positive, HER2 negative, progressive metastatic breast cancer after one or more lines of endocrine therapy (ET) who are initiating a new ET will be enrolled into the study. Patients must have immunohistochemistry (IHC) proven ER positive disease, IHC and/or fluorescence in-situ hybridization (FISH) proven HER2 negative disease, and an ECOG performance status of 0-2. Patients with brain metastases only or those who are progressing on fulvestrant are not eligible for the study.
  Interventions: Other: Blood collection

INTERVENTIONS:
Other: Blood collection — Patients will have blood drawn for circulating tumor cell (CTC) endocrine therapy index (CTC-ETI) calculation at baseline (within 30 days prior to the initiation of endocrine therapy) and then subsequently 1, 2, 3 and up 12 months after the initiation of therapy, or at the time of disease progression, whichever occurs first.

SUMMARY:
Utilizing CellSearch® technology, the ability to both enumerate and reliably and reproducibly characterize circulating tumor cells (CTC) for tumor markers that predict endocrine sensitivity (estrogen receptor [ER] and Bcl-2) and resistance (HER2 and Ki67) has been demonstrated. An algorithm for a CTC-Endocrine Therapy Index (CTC-ETI) has been constructed that can be calculated for each patient using the CTC enumeration and marker results. The primary goal of this study is to determine a CTC-ETI in ER positive, HER2 negative metastatic breast cancer patients before the initiation of a new endocrine therapy for the identification of patients that will progress rapidly.

DETAILED DESCRIPTION:
Patients with estrogen receptor (ER) positive metastatic breast cancer (MBC) starting their first line of endocrine therapy (ET) only have a 30-50% chance of receiving clinical benefit. For the other 50-70% of patients, ET is ineffective and these patients should probably be treated with chemotherapy, as is done for ER negative patients. More importantly, in nearly every clinical trial of ET in ER positive, MBC patients, between 15-30% of enrolled patients progress in the first 2-3 months, regardless of whether they are receiving first or later lines of ET. Currently there is no validated method to identify which ER positive MBC patients will be refractory to ET. Therefore, almost all ER positive patients are treated with serial endocrine therapies before switching to chemotherapy. The investigators propose that a subset of these patients would be better served with chemotherapy, in spite of its increased toxicity profile, rather than delaying chemotherapy during a several month trial of ineffective, albeit less toxic, ET.

To try and predict benefit from or resistance to ET, an index (the CTC-ETI) has been created that takes into account the number of CTC (which is prognostic) as well as the phenotype of the CTC, based on the hypothesis that relative levels of ER and Bcl-2 (high=benefit) and HER2 and Ki67 (high=resistance) are predictive of ET responsiveness or resistance. Although the preliminary data demonstrate the ability to detect, enumerate, and characterize CTC utilizing the CellSearch® System, the purpose of the current study is to establish proof of principle that these 4 markers can be used to generate a CTC-ETI which can be performed at baseline from patients enrolled at different centers, and that baseline CTC-ETI predicts relative outcome for patients with ER positive MBC starting a new ET, and can be monitored in such patients during ET. Successful completion of this study will set the stage for a larger, definitive study designed to demonstrate the clinical utility of a "refined" CTC-ETI in patients with ER positive, HER2 negative MBC.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Women who are 18 years or older.
* Patients must have estrogen receptor (ER) positive, HER2 negative metastatic breast cancer (MBC) with at least one non-irradiated distant site of metastasis.
* ECOG performance status of 0-2.
* Patients must have currently progressive metastatic disease according to RECIST v1.1 criteria, AND

  * They have progressed on at least one previous line of endocrine therapy (ET) for their metastatic disease (but are not currently progressing on fulvestrant), OR;
  * They show evidence of disease progression during or within 12 months of the end of adjuvant ET.
* Patient is about to start a new line of ET for their metastatic disease
* Patient is willing and able to undergo standard of care imaging studies (same imaging/staging modality being used at each evaluation), which are anticipated to be performed prior to the initiation of therapy and subsequently every 3 months.
* Patient agrees to the collection and testing of their blood and is willing and able to provide approximately 40mL blood draw(s) at:

  * Baseline (prior to the initiation of new ET), and;
  * Subsequently at 1, 2, 3 and 12 months after the initiation of therapy, and/or;
  * Time of disease progression.

Exclusion Criteria:

* Patients with local regional recurrence only or brain only metastasis.
* Patients who are progressing on current fulvestrant therapy (patients who have had fulvestrant therapy in the past and were subsequently treated with other therapies or those who are starting fulvestrant as their next line of ET are eligible for the study).
* Patients who are or will be taking other unapproved (i.e. not cleared/approved by the FDA) anti-neoplastic therapies concurrently are not eligible (exception: ET with everolimus is acceptable).
* Patients with concomitant malignancies or previous malignancies within the last 5 years, with exception of adequately treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix.
* Unable to provide informed consent or high risk that patient may not comply with protocol requirements (i.e. due to health and/or participation in other research studies).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients 18 years or older with estrogen receptor (ER) positive, HER2 negative, progressive metastatic breast cancer (MBC) after one or more lines of endocrine therapy (ET) who are initiating a new ET will be enrolled into the study. Patients must have immunohistochemistry (IHC) proven ER positive disease, IHC and/or fluorescence in-situ hybridization (FISH) proven HER2 negative disease, and an ECOG performance status of 0-2. Patients with brain metastases only or those who are progressing on fulvestrant are not eligible for the study.
Sampling Method: Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2016-11-10 (Actual); Study Completion 2016-11-10 (Actual)

PRIMARY OUTCOMES:
Rapid Disease Progression | Within 3 months after initiation of a new line of enrocrine therapy
  Within 30 days prior to the initiation of therapy, chest & abdomen body imaging (computed tomography [CT], or magnetic resonance imaging [MRI] scanning) plus bone scintigraphic imaging (bone scans or PET scans) or PET-CT scans which encompass both will be performed to identify target and non-target lesions that will be followed with the same imaging techniques 3 months after the initiation of therapy. Objective tumor response will be determined using RECIST v1.1 criteria. Rapid disease progression will be defined as disease progression according to RECIST v1.1 criteria or death due to metastatic breast cancer within 3 months of starting a new ET.

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to 12 months after initiation of therapy
  Within 30 days prior to the initiation of of a new line of endocrine therapy (ET), chest & abdomen body imaging (computed tomography [CT], or magnetic resonance imagine [MRI] scanning) plus bone scintigraphic imaging (bone scans or PET scans) or PET-CT scans which encompass both will be performed to identify target and non-target lesions that will be followed with the same imaging techniques 3 months, 6 months, 9 months, and up to 12 months after the initiation of therapy. Objective tumor response will be determined using RECIST v1.1 criteria. Progression Free Survival (PFS) will be measured as the time from the date of starting ET until the date of first documentation of progressive disease according to RECIST v1.1 criteria or death due to any cause. In the absence of these events, PFS will be censored at the date of the last objective disease assessment (up to a maximum of 12 months after the initiation of ET).

OTHER OUTCOMES:
Biomarker correlations | End of study (up to 12 months after enrollment of final patient)
  Correlate the status of the biomarkers on baseline circulating tumor cells (CTC) with the status of the same biomarkers in primary and/or metastatic tissue collected from the patients.
Analytic Validity | Baseline blood draw (within 30 days prior to the initiation of therapy)
  Demonstrate that the circulating tumor cell (CTC) endocrine therapy index (CTC-ETI) can be accurately determined at initiation of a new endocrine therapy (baseline) in patients with ER positive, HER2 negative metastatic breast cancer in multiple centers across North America. Baseline blood sample will be evaluated for the following:
  * successful calculation of CTC-ETI;
  * successful enumeration of CTC in the four aliquots;
  * successful determination of CTC Bio-Score for all 4 markers when the average number of cells is ≥5 CTC/7.5mL of blood.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel F Hayes, M.D., Principal Investigator — University of Michigan Rogel Cancer Center; Costanza Paoletti, M.D., Principal Investigator — University of Michigan Rogel Cancer Center
Locations (20):
- United States (18):
  - Arizona Oncology Associates, Phoenix, Arizona
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Dana-Faber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Minnesota Oncology Hematology, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - New York Oncology Hematology, New York, New York
  - Waverly Hematology Oncology, Cary, North Carolina
  - Duke University, Durham, North Carolina
  - Northwest Cancer Specialists, Portland, Oregon
  - Abramson Cancer Center, University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Texas Oncology - Baylor, Dallas, Texas
  - Texas Oncology, Houston, Texas
- Canada (2):
  - Mt. Sinai Hosp., Marvette Koffler Breast Center, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Background] Paoletti C, Connelly MC, Chianese D, et al. Multi-parameter molecular characterization of circulating tumor cells (CTC): Development of a CTC-Endocrine Therapy Index (CTC-ETI). Proc Am Assoc Cancer Res, Abstract 4154, 2011.
- [Background] Paoletti C, Connelly M, Chianese D, et al. Development of Circulating Tumor Cell-Endocrine Therapy Index in Metastaic Breast Cancer Patients. Cancer Research 71(24 Suppl):451 (Abs. P4-07-16), 2011.